CLINICAL TRIAL: NCT06384768
Title: The Effect of Video Training on Pre-Pregnancy Fear of Birth in Male Partners: A Randomized Controlled Study
Brief Title: Video Training on Pre-Pregnancy Fear of Birth in Male Partners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Elif Balkan, PhD Student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EBIst; 1919B012104428 (Other Grant/Funding Number: TUBITAK)
Record Dates: First submitted 2024-04-23; First posted 2024-04-25 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Fear of Childbirth
Keywords: fear; birth; pregnancy; male; online support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The arm that which was given an online video training
  Interventions: Other: Video training
- Control (No Intervention): No intervention was applied

INTERVENTIONS:
Other: Video training — A 4 week support program consist of videos for fear of childbirth
  Arms: Intervention

SUMMARY:
This study aimed to evaluate the effect of an online video training on fears surrounding childbirth given to male partners before the pregnancy of their spouses. The study conducted with 43 male (22 intervention; 21 control) participants. Participants were divided into intervention and control groups. The intervention group was given video training on pregnancy and the birth process. "Descriptive Information Form" and the "Male-Childbirth Fear Prior to Pregnancy Scale" was used for data collection. Before the intervention, it was found that the fear level of childbirth was low. The video training given to male partners before the pregnancy of their spouses diminished the fear of birth but did not create a significant difference. These findings support long-term training that includes video tutorials for parents before birth. Interactive, participatory birth preparation training is likely to enhance the training's appeal for male partners.

ELIGIBILITY:
Inclusion Criteria:

(i) must be married (ii) must be male gender (iii) must participate voluntarily

Exclusion Criteria:

(i) to have a spouse who had been previously pregnant or having a living child.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Men who have non-pregnant wives.
Enrollment: 43 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Fear of Childbirth | From enrollment to the end of the training at 4 weeks
  Pre-pregnancy fear of childbirth

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Ethical reasons